CLINICAL TRIAL: NCT06198556
Title: A Single Center, Single Arm, Open, Fixed Sequence Study on the Pharmacokinetic Effects of Rifampicin on Oral Administration of HRS-1167 in Healthy Subjects
Brief Title: Effect of Rifampicin on the Pharmacokinetics of HRS-1167 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1167-102
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: Compare the pharmacokinetic effects of Rifampicin on HRS-1167 in healthy subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-1167 with rifampicin (Experimental)
  Interventions: Drug: HRS-1167 tablets; rifampicin

INTERVENTIONS:
Drug: HRS-1167 tablets; rifampicin — HRS-1167 tablets single oral dose of HRS-1167 or co-administered with rifampicin.

SUMMARY:
The primary objective of the study is to evaluate the effect of rifampicin on pharmacokinetics of healthy adult subjects after oral administration of HRS-1167 tablets. The secondary objective of the study is to evaluate the safety of HRS-1167 alone and when co-administered with rifampicin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects aged 18 to 50 years old at the date of signing the informed consent;
2. Weight ≥ 50 kg for male, weight ≥ 45 kg for female, body mass index (BMI): 19~28 kg/m2 (including critical value);
3. Female patients of childbearing age who are not surgically sterilized and male patients whose partners are women of childbearing age must use highly effective contraceptive measures from the signing of the informed consent form to 6 months after the last dose of HRS-1167; female patients of childbearing age who are not surgically sterilized must have a negative serum HCG test within 7 days before the first dose, and must be non-lactating;
4. Be able to communicate well with the investigators and understand and comply with the requirements in this study.

Exclusion Criteria:

1. History of or currently suffering from any serious clinical diseases such as diseases in circulatory system, endocrine system, nervous system, digestive system, respiratory system, genitourinary system, hematology, immunology, psychiatry, and metabolic abnormalities, or any other diseases may interfere with the test results
2. Any surgery within 6 months before screening, or plan to perform surgery during the study period, or who have previously undergone any surgery that affects gastrointestinal absorption (including gastrectomy, bowel resection, gastric reduction surgery, etc.);
3. Those who donate blood or other reasons of bleeding cause the total loss of blood more than 400mL, or receive blood transfusions, or used blood products within 3 months before screening;
4. Allergic constitution, including severe drug allergy or history of drug allergy; Have allergic history to HRS-1167 tablets, rifampicin, rifamycin or their accessories;
5. Frequent use of sedatives, sleeping pills or other addictive drugs; History of drug abuse within 1 year prior to screening; Positive for urine drug abuse screening test;
6. Have taken hepatotoxic drugs (such as dapsone, erythromycin, fluconazole, ketoconazole, rifampicin, etc.) for a long time (continuous administration for more than 7 days) within 6 months before screening;
7. Those who have participated in any clinical trials and taken study drugs within 3 months before the first administration;
8. Have used any drugs that effect enzyme activity within 28 days prior to taking the study drug;
9. Used any prescription drugs and Chinese medicines within one month before the first administration; Have used any over-the-counter drugs (OTC) or food supplements (including vitamins and calcium tablets, etc.) within 2 weeks prior to the first administration;
10. Those who smoke more 5 cigarettes per day in the 3 months before screening or those who do not agree to quit smoking during the test, or those who are positive for urine nicotinic screen;
11. Alcohol abuse in the 6 months prior to screening, with an average weekly intake of more than 14units of alcohol (1 unit = 285 mL of beer, 25 mL of spirits, or 100 mL of wine), and those who cannot abstain from alcohol during the trial, or those who have a positive alcohol breath screening;
12. The results of vital signs, physical examination, 12-lead electrocardiogram, B-ultrasound, chest X-ray, blood-routine examination, blood biochemistry, urine-routine examination, and coagulation function are abnormal during the screening and judged by the research doctor as clinically significant.
13. Those who are positive for HBsAg, HCV antibody, syphilis antibody and HIV antibody.
14. From 48 hours before taking the study drug to the end of the study, subjects have xanthine-rich beverages (chocolate, coffee, tea, etc.) or food; From 7 days before taking the study drug to the end of the study, subjects have; Can't comply with the unified dietary arrangement or have special requirements for diet;
15. Who have blood phobia and faint with acupuncture; or those with poor vascular conditions, inability to embed needles or inability to tolerate venipuncture;
16. Pregnant and lactating women;
17. Subjects who are judged by researchers to be unsuitable for participating in this test.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of HRS1167: Cmax | Based on pre-dose, 0-72 hours post-dose sampling times
Pharmacokinetics parameters of HRS1167: AUC0-t | Based on pre-dose, 0-72 hours post-dose sampling times
Pharmacokinetics parameters of HRS1167: AUC0-inf | Based on pre-dose, 0-72 hours post-dose sampling times

SECONDARY OUTCOMES:
Pharmacokinetics parameters of HRS1167: Tmax | Based on pre-dose, 0-72 hours post-dose sampling times
Pharmacokinetics parameters of HRS1167: t1/2 | Based on pre-dose, 0-72 hours post-dose sampling times
Pharmacokinetics parameters of HRS1167: λz | Based on pre-dose, 0-72 hours post-dose sampling times
Pharmacokinetics parameters of HRS1167: AUC_%Extrap | Based on pre-dose, 0-72 hours post-dose sampling times
Incidence and severity of adverse events/serious adverse events (base on CTCAE 5.0) | From Day 1 to Day 24 after dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided